CLINICAL TRIAL: NCT05817396
Title: Take Care! - Dissemination Von Bewegungsbezogener Gesundheitskompetenz in Der Pflegeausbildung
Brief Title: Dissemination of Physical Activity-related Health Competence in Vocational Education of Nursing Care
Acronym: TakeCare!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Bayerisches Staatsministerium für Gesundheit und Pflege (Bavarian Federal State) (Unknown); Kaufmännische Krankenkasse KKH (Health Insurance) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Chair Lead, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K1-2497-GLB-21-V1
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Physical Activity; Exercise; Education; Nursing; Competence
Keywords: Nursing Students; Physical-Activity related Health Competence; Implementation; Dissemination; Co-creation; Intervention Development
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster-Randomized Controled Trial (cRCT) with 16 schools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cooperative Planning for Promoting PAHCO (Experimental): Participatively developed intervention concept by means of cooperative planning (Rütten, 1997) to promote physical activity-related health competence (PAHCO): A separate cooperative planning process will take place in each of the four schools in this study arm from April to November 2023. Within the framework of these processes, suitable interventions tailored to the target group and the school will be developed for the implementation of the curriculum content "PAHCO" with the participation of actors from science and practice (e.g., teachers, nursing students of the schools). The developed interventions will be implemented from December 2023 under the responsibility of the actors in the schools.
  Interventions: Behavioral: Promotion of Physical Activity-related Health Competence (PAHCO)
- Expert-Based Intervention for Promoting PAHCO Delivered by External Physical Activity Specialists (Experimental): Expert-based intervention concept with external physical activity specialists to promote physical activity-related health competence (PAHCO). We will develop a specific intervention concept for the implementation of the curriculum content "PAHCO" at nursing schools in Bavaria from April to November 2023. Currently (March 2022), it is planned that the intervention will comprise 12 sessions with a duration of 45 or 90 minutes. The entire intervention will be specified during the different steps of intervention mapping (i.e., needs assessment, goal formulation, screening evidence-based intervention content). Physical activity specialists (e.g. sports scientists, physiotherapists) will be trained to implement this expert-based intervention concept from December 2023 to March 2024.
  Interventions: Behavioral: Promotion of Physical Activity-related Health Competence (PAHCO)
- Expert-Based Intervention for Promoting PAHCO Delivered by Teachers (Experimental): Expert-based intervention concept with teachers as multipliers to promote physical activity-related health competence (PAHCO). We will develop a specific intervention concept for the implementation of the curriculum content "PAHCO" at nursing schools in Bavaria from April to November 2023. Currently (March 2022), it is planned that the intervention will comprise 12 sessions with a duration of 45 or 90 minutes. The entire intervention will be specified during the different steps of intervention mapping (i.e., needs assessment, goal formulation, screening evidence-based intervention content). Teachers of the participating nursing schools of this study arm will be trained to implement this expert-based intervention concept in their school from December 2023 to March 2024.
  Interventions: Behavioral: Promotion of Physical Activity-related Health Competence (PAHCO)
- Regular Education and Health Promotion (No Intervention): No systematic intervention concept: In the schools of this study arm, there is no systematic and scientifically supported intervention for the implementation of the curriculum content "PAHCO".

INTERVENTIONS:
Behavioral: Promotion of Physical Activity-related Health Competence (PAHCO) — Intervention for the curriculum content "PAHCO" at nursing schools in Bavaria
  Arms: Cooperative Planning for Promoting PAHCO; Expert-Based Intervention for Promoting PAHCO Delivered by External Physical Activity Specialists; Expert-Based Intervention for Promoting PAHCO Delivered by Teachers

SUMMARY:
The "TakeCare!" study addresses the problem that vocational students of nursing care cope with great physical and psychological demands during their daily routines. To meet these demands, the Bavarian curriculum for generalist nurses has adopted the promotion of physical activity-related health competence (PAHCO) for vocational students. However, it must be assumed that the concept has not yet been adopted comprehensively across the Bavarian nursing landscape. Therefore, the "TakeCare!" study tackles the question of how PAHCO can be implemented most appropriately in Bavarian nursing schools. Drawing on experiences from the project PArC-AVE, three different dissemination approaches will being tested and compared with a control group. A total of 16 nursing schools from different regions of Bavaria will be assigned to four different study arms (cluster-randomized design). In the long term, the project aims to derive recommendations for all nursing schools in Bavaria.

ELIGIBILITY:
Inclusion Criteria (School/Cluster Level):

* Private or Local Sponsorship
* Location in Bavaria
* Schools with 33-64 students in the first cohort (i.e., two or three classes per cohort)
* School director providing informed written consent by March 1st 2023

Inclusion Criteria (Student Level):

* Informed written consent to participate (or their legal guardians, if aged under 18 years)
* Part of the first education year (in cohort 2023/2024)

Exclusion Criteria:

-if any of the criteria mentioned above is not given

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity-related Health Competence (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  Physical Activity-related Health Competence (PAHCO) Questionnaire (Carl et al., 2020); higher percentage scores (0 min, 100 max) indicate a better outcome
Psychological Movement Quality (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  Physical Activity Enjoyment Scale (PACES; Jekauc et al., 2020); higher scores (16 min, 80 max) indicate a better outcome
Quality Physical Activity (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  The outcome is a relational aggregate index between leisure time physical activity and occupational physical activity; higher values (i.e., higher leisure time physical activity relative to occupational physical activity) indicate a better outcome; Leisure time physical activity via BSA Questionnaire (Fuchs et al., 2015); Occupational sitting and physical activity questionnaire (OSPAQ; Chau et al., 2012)
Physical Activity-related Health Competence (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  Physical Activity-related Health Competence (PAHCO) Questionnaire (Carl et al., 2020); higher percentage scores (0 min, 100 max) indicate a better outcome
Psychological Movement Quality (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  Physical Activity Enjoyment Scale (PACES; Jekauc et al., 2020); higher scores (16 min, 80 max) indicate a better outcome
Quality Physical Activity (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  The outcome is a relational aggregate index between leisure time physical activity and occupational physical activity; higher values (i.e., higher leisure time physical activity relative to occupational physical activity) indicate a better outcome; Leisure time physical activity via BSA Questionnaire (Fuchs et al., 2015); Occupational sitting and physical activity questionnaire (OSPAQ; Chau et al., 2012)

SECONDARY OUTCOMES:
General Health Status (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  Single-Item (#1) of the Short-Form-Health-Survey (SF-12; Morfeld et al., 2011); after inversion, higher values (0 min, 4 max) will indicate a better outcome
Work Ability (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  Work Ability Index, short form (WAI-r; Hetzel et al., 2014); higher values (5 min, 36 max) will indicate a better outcome
Musculoskeletal Complaints (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  Ten items (neck/cervical spine, shoulder joints, ellbow/lower arms, hands, thoracic spine, lower back, hip joints/thighs, knee joints, lower legs, feet) of the Nordic Musculosceletal Questionnaire (NMQ; Bundesanstalt für Arbeitsschutz und Arbeitsmedizin, 2021); lower values will indicate a better outcome
Physical Job Stress in Nursing (Short Term) | Change from baseline (T0) to post-intervention (T2; i.e., one year after the baseline)
  Self-developed questionnaire for the physical job stress in nursing; instrument (at its early stage) currently comprises 30 items, will undergo psychometric validation at baseline (T0), lower values (min 0, max 4 for each item) will indicate a better outcome
General Health Status (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  Single-Item (#1) of the Short-Form-Health-Survey (SF-12; Morfeld et al., 2011); after inversion, higher values (0 min, 4 max) will indicate a better outcome
Work Ability (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  Work Ability Index, short form (WAI-r; Hetzel et al., 2014); higher values (5 min, 36 max) will indicate a better outcome
Musculoskeletal Complaints (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  Ten items (neck/cervical spine, shoulder joints, ellbow/lower arms, hands, thoracic spine, lower back, hip joints/thighs, knee joints, lower legs, feet) of the Nordic Musculosceletal Questionnaire (NMQ; Bundesanstalt für Arbeitsschutz und Arbeitsmedizin, 2021); lower values will indicate a better outcome
Physical Job Stress in Nursing (Medium Term) | Change from baseline (T0) to follow-up (T3; i.e., one year after the end of the intervention, two years after the baseline)
  Self-developed questionnaire for the physical job stress in nursing; instrument (at its early stage) currently comprises 30 items, will undergo psychometric validation at baseline (T0), lower values (min 0, max 4 for each item) will indicate a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Alexander University Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenz E, Grune E, Popp J, Pfeifer K, Carl J. Focus group-supported development and psychometric exploration of an instrument to assess perceived physical exertion in nursing students. BMC Nurs. 2024 Dec 30;23(1):957. doi: 10.1186/s12912-024-02639-9. PMID 39736619
- [Derived] Carl J, Grune E, Popp J, Hartung V, Pfeifer K. Implementation and dissemination of physical activity-related health competence in vocational nursing training: study protocol for a cluster-randomized controlled intervention trial. Trials. 2024 May 15;25(1):322. doi: 10.1186/s13063-024-08153-2. PMID 38750590
- See also: Project description on university website — https://www.sport.fau.eu/das-institut/forschung/bewegung-und-gesundheit/forschungsprojekte/takecare/